CLINICAL TRIAL: NCT02465047
Title: Stress and Seizures - Can a Brief Self-help Book Help?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STH17299
Record Dates: First submitted 2015-04-17; First posted 2015-06-08 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Epilepsy; Dissociative Seizures
MeSH Terms: conditions — Epilepsy; Psychogenic Nonepileptic Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-help booklet (Experimental): The intervention consists of a brief A5 self-help stress management booklet with an audio Compact Disk.
  Interventions: Other: Self-help booklet
- Delayed Intervention (No Intervention): Participants do not receive the intervention until one month after the initial assessment.

INTERVENTIONS:
Other: Self-help booklet — See Arm/Group Description
  Arms: Self-help booklet

SUMMARY:
Background: Epilepsy and nonepileptic attack disorder (NEAD) are chronic conditions that cause many patients to experience a great degree of stress in their everyday lives. Patients have also reported stress as the commonest trigger of their seizures, and animal studies suggest that stress can make seizures worse. A self-help intervention that would help people manage the stress they experience could therefore improve their quality of life and have positive effects on the frequency of their seizures.

Research Question: The study evaluates whether a self-help intervention in the form of a brief booklet can improve the quality of life and reduce the levels of stress of people who experience seizures. In addition, the study will explore the associations between seizure severity and frequency, physiological and self-reported stress, and anxiety and depression.

Design: The researchers are recruiting patients attending the Outpatient Neurology Clinic at the Royal Hallamshire Hospital and measure their quality of life and stress levels before, one month and two months after they have been given the self-help stress reduction booklet. The researchers will measure the changes in quality of life and stress levels using questionnaires and saliva samples.

DETAILED DESCRIPTION:
The study is a prospective randomised controlled trial. Patients are randomised to two groups, (1) an immediate intervention group that receives the self-help intervention immediately after recruitment, and (2) a delayed intervention group which receives the intervention at one-month follow-up. Patients are assessed at baseline, at one-month and at two-month follow-up.

Patients attending the neurology outpatient clinic with a confirmed diagnosis of either epilepsy or NEAD are invited to take part in the study. The diagnosis is based on a clinical judgement of a consultant neurologist. Information concerning the purposes and procedures of the study is sent to patients at least 48 hours in advance of their appointment in the neurology outpatient clinic.

Potential participants are screened for their suitability to take part in the study when they come to the neurology clinic. This is based on the exclusion/inclusion criteria and the patients' motivation to participate, which is assessed by five questions asking about the relevance of stress to their lives and to their seizure experiences as well as their interest in participating. Suitable participants have an opportunity to discuss any questions which have arisen from reading the patients information sheet with a member of the research team. Patients willing to take part in the project sign a consent form and complete a set of baseline questionnaires at the time of their hospital appointment with the neurologist, assessing their demographic characteristics, quality of life, stress levels, anxiety, depression, seizure frequency and severity, and their tendency to self-affirm spontaneously. As part of the baseline assessment, patients are also asked to provide two salivary samples the following day (one at 9am in the morning, one at 10pm in the evening) for a measure of baseline levels of salivary cortisol as a marker of physiological stress. Patients complete a seizure diary for the duration of the study.

Patients receive treatment according to the random allocation to the immediate or delayed intervention groups. Patients in the immediate intervention group are provided with a booklet containing the self-help materials as soon as they have provided baseline data and before they leave the hospital on the day of recruitment. They are encouraged to read and work through the booklet over the following week and the researcher contacts them by telephone one week after the baseline assessment, in order to check their progress and to obtain feedback on the booklet, provided they had previously consented to being contacted by telephone.

The first follow-up is arranged for both groups at one month after the initial assessment. Subjects are contacted by post. The follow-up assessment involves completing the quality of life, stress, anxiety, depression, and seizure severity questionnaires, submitting the seizure diary for the past month and providing two saliva samples, one in the morning and one in the evening. Patients in the delayed intervention group also receive the self-help intervention booklet as part of the first follow-up assessment and are encouraged to use the booklet in an accompanying letter. Patients in the delayed intervention group are further contacted by telephone one week after receiving the booklet and asked to provide feedback on their progress and on the booklet itself.

Both groups are then contacted again by letter (or telephone) for a final follow-up two months after the initial assessment. Participants are asked to complete the quality of life, stress, anxiety, depression, and seizure severity questionnaires, to submit their seizure diaries and to provide two final saliva samples, one in the morning and one in the evening.

ELIGIBILITY:
Inclusion Criteria:

* Clinically firm diagnosis of epilepsy (and no additional NEAD) or NEAD (and no additional epilepsy)
* Over the age of 16 years
* Able to complete the self-report questionnaires and diary measure without help
* Able to give informed consent

Exclusion Criteria:

* Patients likely to have mixed seizure disorders (epilepsy and NEAD)
* People who are unable to give informed consent
* People who are unable to complete the self-report questionnaires and diary measure unaided
* People who have not experienced a seizure within the last 12 months
* People whose diagnosis remains uncertain

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Health-related Quality of Life | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Markus Reuber, Professor, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom